CLINICAL TRIAL: NCT06917300
Title: Virtual Reality as a Digital Premed to Alleviate Pain and Anxiety Preoperatively in Patients Undergoing Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Lodz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Supportive Care
Other Study IDs: RNN/02/24/KE
Record Dates: First submitted 2025-02-16; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Anxiety and Fear; Pain, Postoperative; Stress
MeSH Terms: conditions — Anxiety Disorders; Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual Reality (VR) Group - Hospital Environment Exposure (Experimental): This VR group will be exposed to a unified 15-minute VR video via phone using a VR device and goggles after receiving routine standard care. A 360˚ video with an immersive audio-visual environment describing pre-operative and post-operative experience on the day of the surgery will be provided, by which they can get accustomed to the environment and procedures associated with the surgery.
  Interventions: Device: Virtual Reality
- Virtual Reality (VR) Group - Nature Scenery Exposure (Active Comparator): Patients within this group will be provided with standard routine care followed by VR exposure to an immersive environment (i.e., natural scenery, urban parks, tropical beaches, forests) with background music using a commercially available application (i.e., Nature Treks) through a head-mounted display (HMD) and headsets
  Interventions: Device: Virtual Reality
- Standard Care (Control) Group (No Intervention): The standard group, in which patients will only receive standard care and be provided with routine descriptions of the pre-operative experience, where a surgeon will explain to them what the pre-operative experience would entail.

INTERVENTIONS:
Device: Virtual Reality — The VR group will be exposed to a unified 15-minute VR video via phone using a VR device and goggles after receiving routine standard care. A 360˚ video with an immersive audio-visual environment describing pre-operative and post-operative experience on the day of the surgery will be provided, by which they can get accustomed to the environment and procedures associated with the surgery. Background audio will be provided through headsets, and the video will be directed by a neurosurgeon filmed using a Max 360 action VR camera. In the video, actors, neurosurgeons, and nurses will re-enact a typical day for a mock patient undergoing surgery, plus routine post-operative care, including the post-operative immediate recovery room and rehabilitation care by neurosurgeons, psychologists, and physiotherapists in the ward. Patients are allowed to move around freely so that they can experience all aspects of the virtual space, and are encouraged to ask questions at the end.
  Arms: Virtual Reality (VR) Group - Hospital Environment Exposure; Virtual Reality (VR) Group - Nature Scenery Exposure

SUMMARY:
The aim of this research study is to evaluate the impact of immersive VR exposure on preoperative anxiety and pain. Additionally, to assess whether VR intervention would significantly alleviate pain and anxiety levels of patients undergoing complex spinal surgeries. Investigators hypothesize that the application of pre-operative VR-based intervention will alleviate anxiety and pain both pre- and post-operatively when it is used as treatment to complement standard care compared to standard routine care alone, and that it may lead to better outcomes and higher satisfaction in patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 25-70 years old, undergoing an elective spinal surgery.
* Patient's admission prior to surgery day (at least 1 day).
* Expected hospital stay - 2 days.
* Capable of providing informed consent and participate in the study follow-up questionnaire.
* Patients speak Polish.

Exclusion Criteria:

* Congestive heart failure, hypertension and anti-hypertensive medications
* Adrenal insufficiency
* Alcohol addiction (evaluated by CAGE/AUDIT) and substance addiction (evaluated by DUDIT)
* Cognitive impairment (evaluated by MMSE, MoCA)
* Cerebrovascular diseases, ophthalmological diseases (strabismus, diplopia, retina degeneration, glaucoma), neurological conditions (epilepsy or seizure, dementia, vertigo, dizziness, motion sickness) - evaluated by: history taking, examination, vision test (Ishihara test), Simulator Sickness Questionnaire
* Auditory impairment
* Psychiatric illness (schizophrenia, bipolar disorder, psychotic depression) - (evaluated by MINI questionnaire)
* Patients with neuropathic pain
* Use of sedative drugs, anti-depressants, anxiolytics, and anti-epileptic drugs
* Intracranial functional lesions (patients after TBI (Traumatic Brain Injury), cognitive or executive dysfunction)
* Patient with high risk due to major and emergency operations
* Claustrophobia
* GCS < 15

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Stress (STAI-S) and Pain (VAS) | 24 hours postoperatively
  The Primary outcome for this trial is the change in the intensity of pre-operative anxiety measured by the State-Trait Anxiety Inventory (STA-I) scale and pain measured by visual Analogue Scale (VAS). These outcomes will be measured pre-operatively on the day before surgery. Measurements will be made again post-operatively - within 24 hours. Pre-operative and post-operative STAI-S and VAS will be compared for data analysis.

SECONDARY OUTCOMES:
Satisfaction (EVAN-G) and Postoperative Stress (PSS-10) | 24 hours postoperatively
  The Secondary outcome will be the patients' quality of life and satisfaction measured by Evaluation du Vecu de l'Anesthesie Generale (EVAN-G) questionnaire and postoperative stress measured by Perceived Stress Scale PSS-10 within 24 hours and used for data analysis, since the level of satisfaction and the stress caused by thinking time spent at pain can contribute to an increased perception of pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Redwan Rahman Jabbar, Lodz, Łódź Voivodeship, Poland